CLINICAL TRIAL: NCT01162902
Title: Comparison of Vascular Remodeling Between Different Antianginal Medication Evaluated by Noninvasive ECG-gated Fundus Photographic Evaluation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Hyo-Soo, Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABC Trial
Record Dates: First submitted 2010-04-30; First posted 2010-07-15 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Stable Angina
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diltiazem treated group (Experimental): Diltiazem 180mg treated group
  Interventions: Drug: Diltiazem treated group
- Bisoprolol treated group (Active Comparator): Bisoprolol 5mg treated group
  Interventions: Drug: Bisoprolol treated group
- Candesartan treated group (Active Comparator): Candesartan 32mg treated group
  Interventions: Drug: Candesartan treated group

INTERVENTIONS:
Drug: Diltiazem treated group — Diltiazem 180mg for 9 months
  Arms: Diltiazem treated group
Drug: Bisoprolol treated group — Bisoprolol 5mg for 9 months
  Arms: Bisoprolol treated group
Drug: Candesartan treated group — Candesartan 32mg for 9 months
  Arms: Candesartan treated group

SUMMARY:
Treatments for stable angina includes drug therapy such as calcium-channel blocker, beta blocker, and ACEI/ARB. To obtain good prognosis in patients with coronary artery disease,preventing or correcting the progression of atherosclerosis and dyslipidemia is more important than relieving angina symptom. Dysfunction of microvessel is one of the most important factor in patients with coronary artery disease. Recently, we developed the new non-invasive method of evaluating the microvessel in fundus. With this methods, we will compare the effect of each drug (beta blocker, CCB, ARB).

ELIGIBILITY:
Inclusion Criteria:

* Stable angina patients whose coronary lesions is confirmed by angiography or receives PCI
* Unstable Angina/NSTEMI patients who completed PCI for main lesions
* Either systolic > 130mmHg or diastolic > 80mmHg, or patients with anti-hypertensive drugs

Exclusion Criteria:

* STEMI patients within one month
* Variant Angina
* Liver function abnormality or renal failure
* History of Hypersensitivity to testing drugs
* Severe heart failure(NYHA class>3) or uncorrectable hematologic disease
* Woman possible to be pregnant
* Uncontrolled diabetes
* Expected life span < one year

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-01 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Wall to lumen ratio of fundus vessel | baseline, 9 months
  Measurement of change in the ratio of wall thickness to lumen of the fundus vessel from baseline to 9 month follow up

SECONDARY OUTCOMES:
lipid parameter | baseline, 9 months
  Measurement of change in total cholesterol, triglyceride, LDL, small dense LDL, and HDL
Serum markers of inflammation | baseline, 9 months
  CRP
Change of nitrate need | baseline, 1 months, and 3 months
  Measure of change of nitrate need

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea